CLINICAL TRIAL: NCT02063607
Title: The Phase 1a/1b Study of Safety, Pharmacokinetics, Pharmacodynamics of Peglamda (Peginterferon Lamda 1) on Healthy Volunteers and the Preliminary Evaluation of Peglamda and Hepasig (Ribavirin) Treatment's Effects on Chronic Hepatitis C Patients
Brief Title: The Study of Safety, Pharmacokinetics, Pharmacodynamics of Peglamda (Peginterferon Lamda 1) on Healthy Volunteers and the Preliminary Evaluation of Peglamda and Hepasig (Ribavirin) Treatment's Effects on Chronic Hepatitis C Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanogen Pharmaceutical Biotechnology Joint Stock Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NNG01
Record Dates: First submitted 2014-02-11; First posted 2014-02-14 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2014-02

CONDITIONS: Hepatitis C
Keywords: Hepatitis C naive
MeSH Terms: conditions — Hepatitis C | interventions — peginterferon lambda-1a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Peginterferon alfa 2a (Active Comparator): Peginterferon alfa 2a 180 mcg
  Interventions: Biological: Peginterferon lambda
- Peginterferon Lambda (Experimental): Peginterferon Lambda 60,120,180 and 240 mcg
  Interventions: Biological: Peginterferon lambda

INTERVENTIONS:
Biological: Peginterferon lambda

SUMMARY:
This is an open label, dose ranging, phase1a/1b clinical trial to study the safety, Pharmacokinetics and Pharmacodynamics of Peglamda 60, 120, 180 and 240 mcg in healthy volunteers and antiviral activity of once weekly Peglamda administration in combination with daily Ribavirin in Hepatitis C naive patients up to 4 weeks period. The objective of the study to establish safety, PK/PD data on healthy subjects and preliminary efficacy and safety in Hepatitis C naive patients.

ELIGIBILITY:
Inclusion Criteria:

Phase 1a: The subjects who are willing to participate in Phase 1a study must meet ALL of the following inclusion criteria:

1. Volunteers (male and female) between the ages of 18-45
2. Women have a negative pregnancy test result at the time of study.
3. Clinical examination and result laboratory for 7 days before starting the trial must be inside the normal range.
4. Currently not following any treatment regimen (except for using the oral contraceptive).
5. Body mass index is between the range and / or not 25% difference compared to the normal BMI (Appendix 6).
6. Be able to comply with protocol and exchange information effectively with the researchers, agree on the written informed consent to participate in the clinical trial

Phase 1b: Subjects willing to participate into the phase 1b study must meet ALL of the following inclusion criteria:

1. Patients with chronic hepatitis C (male and female).
2. Ages between 18 - 65 years old.
3. Female patient (or female partners of the male patients) with negative pregnancy test results and/or apply effective contraception if still having sex during the study and for 6 months after using the last dose of Ribavirin.
4. No previous treatment with IFN or IFN treatment with rapid viral response or already have completely viral response but leave the treatment early.
5. HCV-RNA levels in serum > 80 IU / mL.
6. The haematological and biochemical (except ALT / AST) parameters must be within normal limits.
7. Body weight in the normal range of 25% difference compared to the normal BMI (Appendix 6)
8. Be able to comply with protocol and exchange information effectively with the researchers, agree on the written informed consent to participate in the clinical trial

Exclusion Criteria:

Phase 1a: Subjects with at least 1 of the following exclusion criteria are considered ineligible to participate in Phase 1a study:

1. With a history of drug abuse, alcohol or drug using within 1 year before taking part in the clinical trial. AUDIT-C scale (WHO) will be used to assess the use of alcohol. The score ≥ 4 in men or ≥ 3 in women are considered as alcoholics.
2. History of depression
3. History of chronic diseases related to the respiratory system, cardiovascular, gastrointestinal, malignant disease affecting to the function of the organ systems. Having any interferon or antiviral therapy within 4 months before the trial
4. Participate in any clinical trial within 3 months prior the testing
5. Use of any drug in the last period of relatively positive test which last approximately 6 times the half-life of the drug.
6. Blood donor with more than 400 mL of blood within 3 months prior the testing
7. Influenza infection or cold symptoms within 2 weeks before the trial
8. Having positive tests of HBV, HCV or HIV
9. Breastfeeding women

Phase 1b: Subjects with at least 1 of the following exclusion criteria are considered ineligible to participate in Phase 1b study:

1. Co-infection with hepatitis B and/or HIV.
2. Hepatic Impairment
3. Cirrhosis
4. Positive tests with antibody of Peginterferon lambda 1 and Peginterferon alpha 2a.
5. History of chronic diseases related to the respiratory system, cardiovascular, gastrointestinal, malignant disease affecting to the function of the organ systems.
6. A history of immune disorders (eg, inflammatory bowel disease, hemorrhagic thrombocythemia, lupus erythematosus, autoimmune hemolytic anemia, autoimmune disease, scleroderma, severe psoriasis, arthritis rheumatoid ...)
7. A history of severe mental illness, especially depression, especially the serious neurological condition determined as depression or serious psychological disorders, suicidal intention, or being hospitalized for mental illness, or having 1 phase of impaired function due to neuropathy.
8. A history of severe epilepsy or using antiepileptic drugs.
9. A history of using anti-cancer agents (including radiation therapy) or immunotherapy (including systematic corticosteroids) within 6 months before using the first testing dose or the patient may be in need of this treatment during the trial
10. History of organ transplants with the presence of the graft function.
11. Evidence of alcohol or drugs abuse within 1 year before the trial. AUDIT scale - C will be used to assess the use of alcohol. The score ≥ 4 in men or ≥ 3 in women are considered as alcoholics
12. History or evidence of severe disease or any other condition based on the investigator assessment that the subject may not be suitable for this study.
13. Breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve (AUC 0-336) | 0, 6, 12, 24, 36, 48, 72, 96, 120, 144, 168, 216, 264 and 336 hours
Percentage of Patients achieving Rapid Virological Response (RVR) | 4 weeks

SECONDARY OUTCOMES:
Number of subjects with incidence of adverse events | 15 days

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Chinh Trong Nguyen, PhD, Principal Investigator — The Military 108 Hospital
Locations (1):
- The Military 108 Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No